CLINICAL TRIAL: NCT04159428
Title: Validation and Evaluation of the French Version of a Hearing Loss Screening Questionnaire in Adults Aged 60 Years Old and More (Hearing Handicap Inventory for the Elderly Screening Version)
Brief Title: Validation and Evaluation of the French Version of a Hearing Loss Screening Questionnaire in Adults Aged 60 Years Old and More
Acronym: VF DEPIST 60
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/15
Record Dates: First submitted 2019-10-30; First posted 2019-11-12 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Hearing Loss
Keywords: hearing loss; screening; elderly; hidden hearing loss; speech in noise audiometry; HHIE-S survey
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Hidden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HHIE-S survey score — First, the patient will fill in the French translation of the HHIE-S questionnaire in the observation book.
  * Secondly, he will perform the audiometry in silence test: for the tonal test in silence, we will test the frequencies 500, 1000, 2000 and 4000 hertz in each ear with pure tone sound. For the vocal in silence test, we will use the dissyllabic lists of words (Fournier's lists) at the intensities of 20, 30, 40, 50 and 60 decibels. This test will be in free-field conditions testing both ears.
  * Thirdly, he will perform the speech in noise audiometry test that consists in repeating sentences pronounced at an equal intensity (60 decibels) while the intensity of the noise is increasing. This test will be in free-field conditions testing both ears.

SUMMARY:
Nowadays in France, there is no organized screening of the hearing loss in the elderly; however, it is a very common disease and simples tests to perform to detect it exist. Lots of studies use surveys to identify deaf people; but physicians often consider them too sensitive and less specific because lots of people were classified into " deaf " people meanwhile they have a subnormal tonal audiogram.

Now, it's known that it corresponds to the "Hidden Hearing Loss" concept: it's defined as an auditive disturbance in a noisy ambiance in people with a normal tonal audiometry; corresponding to infraclinical cochlear lesions. These lesions, if detected early, can be prevented to avoid an audition degradation in time.

The aim of the study is to determinate the values of sensitivity and specificity of the HHIE-S survey translated into French, so it could be used as a screening method of hearing loss in the elderly and as a prevention of cochlear damages.

DETAILED DESCRIPTION:
The HHIE-S survey is one of the more used in studies to screen hearing loss in elderly. It has never been validated in French: that's why investigatosr want to test it on the French population, to determine its performance characteristics (sensitivity and specificity). Secondary, investigators study think that people that have high score on the hear loss screening survey, but a normal tonal audiometry have actually a hidden hearing loss. This corresponds to infraclinical cochlear lesions that we want to reveal thanks to a new audiometric test: an audiometry in a noisy ambiance.

The study will take place in a research audiometric room in the department of ENT in Bordeaux. Patients will fill a medical survey the HHIE-S survey translated into French and perform a tonal audiometry test and after it a " speech in noise " audiometry test (VRB in French).

The duration os study is one unique session of 45 minutes including patient information and consent.

ELIGIBILITY:
Inclusion Criteria:

* are 60 years old and more
* are able to express their consent
* are affiliated to the French social security

Exclusion Criteria:

* have known hearing problem of any kind
* have performed an audiogram within the past 6 months
* have required medical examination for any hearing problem
* have had ear surgery of any kind (except form myringotomy tube during the childhood)
* have mental or physical serious injury(ies), which results an impossibility to fill a survey and perform an audiogram
* are under protection schemes

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French elderly population without hearing problem
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Surdity assessed with tonal audiometric examination | Inclusion (t0)
  Primary outcome measure is the presence of surdity on one or two ears of the patient.
  This Primary outcome will be evaluated with tonal audiometric examination

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No